CLINICAL TRIAL: NCT05353335
Title: Investigating if Nocturnal Blood Pressure Patterns Are Modifiable in Children With Chronic Kidney Disease
Brief Title: Chronotherapy in Children With Chronic Kidney Disease
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: not justified based on recent analyses of non-dipping in children with CKD
Sponsor: Yale University (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); American Heart Association (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: 2000031575; 1K23DK129836-01 (NIH)
Record Dates: First submitted 2022-04-25; First posted 2022-04-29 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-06

CONDITIONS: Chronic Kidney Diseases; Hypertension
MeSH Terms: conditions — Renal Insufficiency, Chronic; Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- nighttime dosing of one anti-hypertensive medication (Experimental): 13 participants will be randomized to nighttime dosing of one anti-hypertensive medication. After 1 week, a repeat ABPM will be obtained. At 1 month from randomization, another ABPM will be obtained. Following this, there will be a 2-week washout period, during which all subjects will be on their usual anti-hypertensive regimen. A repeat ABPM will be obtained after the washout period. Next, the subjects will crossover to the opposite arm and an ABPM will be obtained after 1 week. A final ABPM will be obtained at 1 month after crossover.
  Interventions: Other: Re-timing of anti-hypertensive drug
- remain on their current regimen (Active Comparator): 13 participants will be randomized to remain on their current regimen. After 1 week, a repeat ABPM will be obtained. At 1 month from randomization, another ABPM will be obtained. Following this, there will be a 2-week washout period, during which all subjects will be on their usual anti-hypertensive regimen. A repeat ABPM will be obtained after the washout period. Next, the subjects will crossover to the opposite arm and an ABPM will be obtained after 1 week. A final ABPM will be obtained at 1 month after crossover.
  Interventions: Other: Current regimen

INTERVENTIONS:
Other: Re-timing of anti-hypertensive drug — The intervention will consist of shifting the anti-hypertensive medication from morning/early dose to an evening/later dose
  Arms: nighttime dosing of one anti-hypertensive medication
Other: Current regimen — The participants will begin on their current regimen.
  Arms: remain on their current regimen

SUMMARY:
This is a pilot, crossover trial in which the investigator will determine if retiming of one anti-hypertensive medication from morning to evening can effectuate normal blood pressure dipping patterns in children and adolescents with chronic kidney disease.

DETAILED DESCRIPTION:
Normally blood pressure declines by at least 10% from daytime to nighttime. In children with chronic kidney disease (CKD), often this does not happen (termed "non-dipping"). This study is a pilot, randomized cross-over trial. The main purpose of this study is to investigate whether non-dipping can be modified with retiming of anti-hypertensives in children with CKD. This is important because in adults, non-dipping has been associated with increased cardiovascular disease risk and more rapid progression of kidney disease. Thus, identification of how to modify this in children with CKD, may lead to future randomized controlled trials to evaluate whether chronotherapy improves outcomes in this population, which is at high risk for morbidity and mortality in adulthood.

The primary objective of this study is to determine whether retiming of one anti-hypertensive to the evening will increase nocturnal systolic blood pressure change (%) in children with CKD, hypertension and non-dipping.

The secondary objective of this study is to determine whether retiming of one anti-hypertensive to the evening will increase nocturnal diastolic blood pressure change (%) in children with CKD, hypertension and non-dipping. Another secondary objective is to determine if the proportion of subjects classified as having a non-dipping pattern is significantly lower on evening dosing of anti-hypertensives.

ELIGIBILITY:
Inclusion Criteria:

* Male or female child/adolescent up to 18 years of age with CKD
* estimated glomerular filtration rate (eGFR) of 30 to 90 ml/min/1.73 m2
* diagnosed with hypertension and on a stable dose of anti-hypertensive medication(s) for at least 3 months
* Non-dipping identified on ABPM

Exclusion Criteria:

* history of organ transplantation, oncological disease, or dialysis
* inability to complete 24-hour ABPM or 24-hour urine collection
* Children less than 6 years of age will be excluded, as they often are unable to complete a successful ABPM study (≥ 40 readings, with 1 reading per hour of sleep)
* Currently on diuretic medications.

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2025-04 (Estimated); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Percent change in nocturnal systolic blood pressure in participants administered anti-hypertensive medications at night on Ambulatory blood pressure monitor(ing) (ABPM). | Baseline and Month 1
  Percent change in systolic nocturnal blood pressure will be calculated as : (daytime mean SBP - nighttime mean SBP)/daytime mean SBP x 100 to assess if nocturnal BP dipping can be restored.

SECONDARY OUTCOMES:
Percent change in nocturnal diastolic blood pressure in participants administered anti-hypertensive medications at night on ABPM. | Baseline and Month 1
  Percent change in systolic nocturnal blood pressure will be calculated as: (daytime mean DBP - nighttime mean DBP)/daytime mean DBP x 100 to assess if nocturnal BP dipping can be restored.
Change in proportion of participants with restoration of dipping while on the intervention, defined as <10% systolic or diastolic nocturnal blood pressure change | Baseline and Month 1
  This outcome will assess if the proportion of subjects classified as having a non-dipping pattern is significantly lower on evening dosing of anti-hypertensives. Restoration of dipping would mean that both systolic and diastolic nocturnal blood pressure change are greater than or equal to 10%, after the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Christine Bakhoum, Principal Investigator — Yale University
Locations (1):
- Yale New Haven Children's Hospital/Yale New Haven Health, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: Yes